CLINICAL TRIAL: NCT05799274
Title: Characterizing the Radiochemical and Radiation Safety of RAD301 in Healthy Human Volunteers and Patients With Pancreatic Ductal Adenocarcinoma or Other Solid Tumors
Brief Title: Safety of RAD301 in Healthy Human Volunteers and Patients With Pancreatic Cancer or Other Solid Tumors
Acronym: RAD301
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Radiopharm Theranostics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RAD301.2022-001
Record Dates: First submitted 2023-03-12; First posted 2023-04-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Pancreatic Ductal Adenocarcinoma; Non-small Cell Lung Cancer (NSCLC); Esophageal Squamous Cell Carcinoma; Cervical Cancer; Endometrial Cancer; Ovarian Cancer
Keywords: Pancreatic Ductal Adenocarcinoma; non-small cell lung cancer (NSCLC); esophageal squamous cell carcinoma; cervical cancer; endometrial cancer; ovarian cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Squamous Cell Carcinoma; Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [68Ga]-RAD301 (Experimental): 150 +/- 50 MBq (~4 mCi) single dose administered at Day 1 visit
  Interventions: Drug: RAD301 ([68Ga]-RAD301)

INTERVENTIONS:
Drug: RAD301 ([68Ga]-RAD301) — A single dose of 68Ga-RAD301 of 150 +/- 50 MBq (~4mCi) administered as a slow bolus injection over 2-5 minutes

SUMMARY:
This is a Phase 1a, open label, single dose, extended study of safety and biokinetics of RAD301 in healthy human volunteers and individuals with PDAC or Other Solid Tumors

DETAILED DESCRIPTION:
This will be a Phase 1a, open label, single dose, extended study of safety and biokinetics of RAD301 in healthy human volunteers and individuals with PDAC or Other Solid Tumors. The procedures will be similar in both groups, but there could be more scans in healthy volunteers and fewer in individuals with PDAC or Other Solid Tumors during the same time interval if individuals are intolerant of lying still on an imaging table for long periods of time. All individuals will have vital signs, ECGs, and blood for safety assessments collected before and 2 weeks after a single dose, intravenous (IV) administration of the investigational radiopharmaceutical, RAD301, at a dose of 150 ± 50 MBq (~ 4 mCi). There will be 3 whole body (WB) PET-CT and PET scanning sessions.

The initial WB acquisition should take approximately 10 minutes. A subsequent WB PET-only scan will be performed approximately 45 minutes after the injection. As time passes and less radioactivity is localizable to the distal extremities, the scan length may be decreased from vertex-to-thighs. The duration of each scan may increase to partially compensate for radioactive decay. More than one WB scan may be performed in healthy volunteers during the first imaging session, but only one scan will be required in individuals with PDAC or Other Solid Tumors who are not able to tolerate additional scans. The entire first imaging session will last up to approximately 2 hours. The individuals will then be given a rest period (lunch break) after which the sequence of imaging scans could be repeated.

This second imaging session (WB PET-CT) will be optional and depends on the robustness of the individual and the availability of the clinical scanner. The second imaging session will take place mid-day, after the break, and will last up to 1.5 hours.

There will be a third, or final imaging session (WB PET-CT) at the end of the day for all participants, which will strive to include the time interval after approximately 4 physical half-lives of Gallium-68 (Ga-68). The third imaging session will last up to 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age at the time of informed consent.
2. All participants must be willing and able to give informed consent.
3. For patients with cancer: have a history of histologically or cytologically confirmed PDAC, non-small cell lung cancer (NSCLC), esophageal squamous cell carcinoma, cervical cancer, endometrial cancer, or ovarian cancer and have had a SOC CT or MRI within 12 weeks prior to giving consent that indicates the presence of at least 1 site of new or residual disease. If the SOC CT or MRI has occurred prior to 12 weeks, consultation with the Sponsor must be sought prior to patient enrollment. SOC images must be available for submission to the centralized imaging reader as reference.
4. Screening laboratory values within 30 days prior to administration of the study drug:

   1. WBC ≥ 1200/μL
   2. ANC ≥ 1000/μL
   3. Platelets ≥ 75,000/μL
   4. Hemoglobin ≥ 9.0 g/dL
   5. Creatinine ≤ 1.5 mg/dL
   6. AST/ALT ≤ 3 x ULN for patients with no liver metastases.
   7. AST/ALT ≤ 5 x ULN for patients with liver metastases.
   8. Bilirubin ≤ 1.5 mg/dL except for participants with Gilbert's disease.
5. Patients should have a life expectancy of ≥ 12 weeks as judged by the Investigator.
6. All participants must have baseline pulse oximetry ≥ 95% on room air.
7. Unremarkable ECGs, with PR intervals of less than 200 msec and QTcF intervals (corrected with Frederica's method) of less than 450 msec.
8. Willing to refrain from taking illicit drugs one week prior to PET scanning and through the follow-up phone call on Day 3 (+2 days).
9. Willing to refrain from donating blood for 4 weeks after administration of RAD301.
10. Have not participated in any other research study that requires taking medication within 4 weeks (or 10 half-lives, whichever is shorter) from the time of informed consent to the end of the Imaging and Safety Follow-Up Period. Previous or ongoing participation in another study should be discussed with the Sponsor.

Exclusion Criteria:

1. Participant may not be a member of a vulnerable population defined as participants who are not able to understand the nature of the trial and provide informed consent or who have any medical, psychological or sociological condition that in the opinion of the investigator would interfere with the ability to give consent or interfere with protocol compliance.
2. Women may not be pregnant or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to administration of RAD301.
3. History of an anaphylactic reaction to a protein- or peptide-derived therapeutic or a diagnostic agent.
4. History, physical examination, or clinical laboratory tests suggestive of a condition, disorder, or disease that could adversely affect drug absorption, distribution, metabolism, or elimination of RAD301, including chronic liver or renal failure.
5. Unable to tolerate the study procedures.
6. Patients with brain metastases are eligible as long as there is no requirement for high doses of systemic corticosteroids that could result in immunosuppression (>10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration. An MRI is not required to rule out brain metastases or leptomeningeal metastases
7. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, or interfere with the interpretation of study results.
8. Clinically significant cardiovascular/ cerebrovascular disease defined as cerebral vascular accident, stroke, carotid artery disease transient ischemic attach (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >II) or serious cardiac arrhythmia.
9. Other than the tumor types being studied, a prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast.
10. Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
11. Participants who underwent major surgery within 4 weeks of administration of study drug (not including diagnostic laparoscopy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Radiation dosimetry of RAD301 | 6 hours
  Absorbed radiation dose of RAD301 in critical organs
Radiation dosimetry of RAD301 | 6 hours
  Absorbed radiation dose of RAD301 in tumor lesions
Safety and tolerability of RAD301 | 4 weeks
  The properties, incidence, nature and severity of AEs and SAEs per Common Terminology Criteria for Adverse Events (CTCAE) v5.0

OTHER OUTCOMES:
Concordance between RAD301 PET and CT or MRI | 1 week
  Proportion of metastases correctly identified by RAD301 out of the total number of metastases confirmed by standard of care (SOC) imaging methods, such as computed tomography (CT) or MRI
Concordance between RAD301 PET and CT or MRI | 1 week
  Proportion of cases correctly identified by RAD301 as having no metastasis out of the total number of cases confirmed to have no metastasis by SOC imaging methods, such as CT or MRI
Concordance of RAD301 PET and CT or MRI | 1 week
  Proportion of all cases correctly identified by RAD301, either as having or not having metastasis, out of the total number of cases, as confirmed by SOC imaging methods, such as CT or MRI
Time Activity Curves (TACs) | 6 hours
  Percent of the injected activity vs time for selected organs
Biokinetics of RAD301 | 6 hours
  Time lag between injection and peak conspicuity in PDAC tumor masses

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - United Theranostics, Princeton, New Jersey
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
Single center study